CLINICAL TRIAL: NCT04018313
Title: A Phase 1, Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of Three Formulations of Omalizumab (CT-P39, EU-approved Xolair, and US-licensed Xolair) in Healthy Subjects
Brief Title: To Compare the PK and Safety of Omalizumab (CT-P39, EU-approved Xolair, and US-licensed Xolair) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P39 1.1
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CT-P39 (Part 1) (Experimental): 150 mg/mL, Solution for injection in PFS
  Interventions: Biological: CT-P39
- EU-approved Xolair (Part 1) (Active Comparator): 150 mg/mL, Solution for injection in PFS
  Interventions: Biological: EU-approved Xolair
- CT-P39 (Part 2) (Experimental): 150 mg/mL, Solution for injection in PFS
  Interventions: Biological: CT-P39
- EU-approved Xolair (Part 2) (Active Comparator): 150 mg/mL, Solution for injection in PFS
  Interventions: Biological: EU-approved Xolair
- US-licensed Xolair (Part 2) (Active Comparator): 150 mg/mL, Solution for injection in PFS
  Interventions: Biological: US-licensed Xolair

INTERVENTIONS:
Biological: CT-P39 — 150 mg/mL, Solution for injection in PFS
  Arms: CT-P39 (Part 1)
Biological: EU-approved Xolair — 150 mg/mL, Solution for injection in PFS
  Arms: EU-approved Xolair (Part 1)
Biological: CT-P39 — 150 mg/mL, Solution for injection in PFS
  Arms: CT-P39 (Part 2)
Biological: EU-approved Xolair — 150 mg/mL, Solution for injection in PFS
  Arms: EU-approved Xolair (Part 2)
Biological: US-licensed Xolair — 150 mg/mL, Solution for injection in PFS
  Arms: US-licensed Xolair (Part 2)

SUMMARY:
A Phase 1, Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of Three Formulations of Omalizumab (CT-P39, EU-approved Xolair, and US-licensed Xolair) in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (male or female) between the ages of 18 and 55 years.
* Subject with a body weight of > 40 kg and ≤ 90 kg and a BMI between 18.0 kg/m2 and 32.0 kg/m2(both inclusive).
* Subject with a total IgE level of ≤ 100 IU/mL.

Exclusion Criteria:

* Subject has a medical history and/or current presence of disease including one or more of the allergic reaction.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SungHyun Kim, Study Director — Celltrion
Locations (2):
- Australia (2):
  - Phase 1 unit, Herston, Queensland
  - Phase 1 unit, Adelaide, South Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P39 (Part 1); CT-P39 (Part 2): Healthy subjects were administered single subcutaneous (SC) injection of CT-P39 via pre-filled syringe (PFS).
  CT-P39: 150 mg/mL Solution for injection.
- EU-approved Xolair (Part 1); EU-approved Xolair (Part 2): Healthy subjects were administered single subcutaneous (SC) injection of EU-approved Xolair via pre-filled syringe (PFS).
  EU-approved Xolair: 150 mg/mL Solution for injection.
- US-licensed Xolair (Part 2): Healthy subjects were administered single subcutaneous (SC) injection of US-licensed Xolair via pre-filled syringe (PFS).
  US-licensed Xolair: 150 mg/mL Solution for injection.
Period: Overall Study
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Started | 15 | 15 | 47 | 49 | 50
Completed | 14 | 14 | 46 | 47 | 49
Not Completed | 1 | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: ITT set: all subjects enrolled and randomly assigned to receive a dose of any study drug, regardless of whether or not any study drug was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2) | Total
Number analyzed (Participants) | 15 | 15 | 47 | 49 | 50 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (6.31) | 26.9 (9.11) | 28.2 (8.81) | 32.1 (11.65) | 30.3 (10.09) | 29.6 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 28 | 27 | 30 | 101
  Male | 7 | 7 | 19 | 22 | 20 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 6 | 6 | 8 | 30
  Not Hispanic or Latino | 9 | 7 | 40 | 39 | 39 | 134
  Unknown or Not Reported | 1 | 3 | 1 | 4 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 0 | 3 | 0 | 0 | 0 | 3
  Asian | 0 | 0 | 7 | 6 | 8 | 21
  Black or African American | 1 | 0 | 0 | 3 | 0 | 4
  Australian Aborigine/Torres Strait Islander | 0 | 0 | 1 | 0 | 0 | 1
  Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  White | 12 | 12 | 36 | 38 | 40 | 138
  Other | 2 | 0 | 2 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  Australia | 15 | 15 | 47 | 49 | 50 | 176
Body mass index at screening [Mean (Standard Deviation); unit: kg/m2] | 22.93 (2.525) | 23.65 (2.306) | 23.90 (3.042) | 23.19 (2.864) | 23.71 (2.980) | 23.54 (2.866)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Outcome Measures [AUC0-inf] for Part 2
Description: Area Under the concentration-time Curve from time zero to infinity (AUC0-inf) of CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects (CT-P39 to EU-approved Xolair, CT-P39 to US-licensed Xolair, and EU-approved Xolair to US-licensed Xolair)
Time Frame: up to day 127
Population: PK set: all randomly assigned subjects who receive a complete dose of study drug and provide at least one post-treatment serum concentration above the lower limit of quantification for omalizumab.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 46 | 49 | 50
day*μg/mL | 910.9 (278.57) | 897.7 (270.25) | 926.3 (273.30)
Statistical Analysis 1: Comparison: CT-P39 (Part 2) vs EU-approved Xolair (Part 2); The statistical analysis of the log-transformed primary endpoints was based on an ANCOVA model with treatment as fixed effect and baseline body weight, total IgE level and sex as covariates; Test type: Equivalence — The similarity of PK between CT-P39 versus EU-approved Xolair, CT-P39 versus US-licensed Xolair, and EU-approved Xolair versus US-licensed Xolair was concluded if the 90% confidence intervals (CIs) of the ratios of geometric means of each comparison are entirely contained within 80% to 125% for AUC0-inf, AUC0-last, and Cmax; Ratio of geometric least square means = 105.62, 90% CI 2-sided [95.91 to 116.31]
Statistical Analysis 2: Comparison: CT-P39 (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 98.72, 90% CI 2-sided [89.76 to 108.58]
Statistical Analysis 3: Comparison: EU-approved Xolair (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 93.47, 90% CI 2-sided [85.09 to 102.68]

2. Primary Outcome: Pharmacokinetic Outcome Measures [AUC0-last] for Part 2
Description: Area Under the concentration-time Curve from time zero to the last quantifiable concentration (AUC0-last) of CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects (CT-P39 to EU-approved Xolair, CT-P39 to US-licensed Xolair, and EU-approved Xolair to US-licensed Xolair)
Time Frame: up to day 127
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 47 | 49 | 50
day*μg/mL | 846 (251.87) | 843.8 (248.04) | 850.0 (213.13)
Statistical Analysis 1: Comparison: CT-P39 (Part 2) vs EU-approved Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 104.00, 90% CI 2-sided [94.96 to 113.89]
Statistical Analysis 2: Comparison: CT-P39 (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 99.30, 90% CI 2-sided [90.79 to 108.61]
Statistical Analysis 3: Comparison: EU-approved Xolair (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 95.48, 90% CI 2-sided [87.36 to 104.37]

3. Primary Outcome: Pharmacokinetic Outcome Measures [Cmax] for Part 2
Description: Maximum serum concentration (Cmax) of CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects (CT-P39 to EU-approved Xolair, CT-P39 to US-licensed Xolair, and EU-approved Xolair to US-licensed Xolair)
Time Frame: up to day 127
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 47 | 49 | 50
μg/mL | 20.08 (5.9940) | 18.24 (4.9981) | 19.43 (5.4159)
Statistical Analysis 1: Comparison: CT-P39 (Part 2) vs EU-approved Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 113.14, 90% CI 2-sided [103.15 to 124.11]
Statistical Analysis 2: Comparison: CT-P39 (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 103.88, 90% CI 2-sided [94.83 to 113.80]
Statistical Analysis 3: Comparison: EU-approved Xolair (Part 2) vs US-licensed Xolair (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least square means = 91.82, 90% CI 2-sided [83.87 to 100.52]

4. Secondary Outcome: Pharmacokinetic Outcome Measures [Tmax] for Part 1& Part 2
Description: To assess Time to Cmax (Tmax) of CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: up to day 127
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 15 | 15 | 47 | 49 | 50
day | 7.178 [5.04 to 56.27] | 7.244 [3.00 to 14.17] | 7.098 [2.00 to 14.26] | 7.306 [3.00 to 18.26] | 7.183 [3.00 to 21.17]

5. Secondary Outcome: Pharmacokinetic Outcome Measures [t1/2] for Part 1& Part 2
Description: To assess Terminal half-life (t1/2) of CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: up to day 127
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 15 | 15 | 46 | 49 | 50
day | 29.75 (3.9477) | 28.77 (5.0315) | 29.30 (9.5158) | 27.69 (5.5603) | 28.63 (6.6290)

6. Secondary Outcome: Pharmacodynamics Outcome Measures [Cmin of Free IgE] for Part 1 & Part 2
Description: To assess the minimum observed concentration (Cmin) of Free IgE in CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: up to day 127
Population: PD set: all randomly assigned subjects who receive a complete dose of study drug and have at least one post-treatment free IgE or total IgE concentration above the lower limit of quantification.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 13 | 11 | 31 | 38 | 32
IU/mL | 3.1538 (1.12963) | 3.4613 (1.43457) | 3.5267 (1.45275) | 3.5590 (1.56235) | 3.7002 (1.69613)

7. Secondary Outcome: Pharmacodynamic Outcome Measures [Tmin of Free IgE] for Part 1 & Part 2
Description: To assess the Time to Cmin (Tmin) of Free IgE in CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: Up to day 127
Population: as for outcome 6
Measure: Median (Full Range); unit: day
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 13 | 11 | 31 | 38 | 32
day | 3.000 [0.50 to 10.09] | 5.196 [1.00 to 126.25] | 3.000 [0.25 to 21.21] | 5.051 [0.25 to 70.17] | 3.002 [0.25 to 41.07]

8. Secondary Outcome: Pharmacodynamic Outcome Measures [Cmax of Total IgE] for Part 1 & Part 2
Description: To assess the maximum observed concentration (Cmax) of total IgE in CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: up to day 127
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 15 | 15 | 46 | 49 | 49
IU/mL | 241.5333 (156.50234) | 165.2000 (122.59702) | 245.2391 (223.24856) | 174.2857 (145.17432) | 219.5714 (187.41287)

9. Secondary Outcome: Pharmacodynamic Outcome Measures [Tmax of Total IgE] for Part 1 & Part 2
Description: To assess the Time to Cmax (Tmax) of total IgE in CT-P39, EU-approved Xolair, and US-licensed Xolair in healthy subjects
Time Frame: up to day 127
Population: as for outcome 6
Measure: Median (Full Range); unit: day
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
Number analyzed (Participants) | 15 | 15 | 46 | 49 | 49
day | 28.263 [20.99 to 69.17] | 28.167 [14.19 to 56.10] | 28.191 [3.00 to 70.13] | 28.156 [14.01 to 71.07] | 28.087 [10.18 to 73.07]

ADVERSE EVENTS:
Time Frame: All AEs were collected from the date the ICF was signed and AE reporting continued until the end of the subject's participation in this study (up to Day 127).
Description: Only treatment-emergent adverse events and treatment-emergent serious adverse events were summarized
Groups:
- US-licensed Xolair (Part 2): Healthy subjects were administered single subcutaneous (SC) injection of US-licensed Xolair via pre-filled syringe (PFS).
  US-licensed Xolair: 150 mg/mL, Solution for injection.
Arm/Group | CT-P39 (Part 1) | EU-approved Xolair (Part 1) | CT-P39 (Part 2) | EU-approved Xolair (Part 2) | US-licensed Xolair (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/47 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/47 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 4/15 | 7/15 | 20/47 | 26/49 | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P39 (Part 1) (N=15) | EU-approved Xolair (Part 1) (N=15) | CT-P39 (Part 2) (N=47) | EU-approved Xolair (Part 2) (N=49) | US-licensed Xolair (Part 2) (N=50)
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P39 (Part 1) (N=15) | EU-approved Xolair (Part 1) (N=15) | CT-P39 (Part 2) (N=47) | EU-approved Xolair (Part 2) (N=49) | US-licensed Xolair (Part 2) (N=50)
Nausea (Gastrointestinal disorders) | 0 | 0 | 6 | 2 | 2
Catheter site pain (General disorders) | 1 | 1 | 0 | 1 | 3
Fatigue (General disorders) | 1 | 0 | 3 | 2 | 3
Injection site reaction (General disorders) | 1 | 1 | 8 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 4
Catheter site irritation (General disorders) | 0 | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 4 | 2
Headache (Nervous system disorders) | 1 | 5 | 11 | 10 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A confidentiality and non-disclosure agreement (CDA) was executed between Celltrion, Inc. and some PIs who have participated in publications funded by the sponsor for academic purposes for a period that is more than 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04018313/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04018313/SAP_001.pdf